CLINICAL TRIAL: NCT02724423
Title: An Open-Label, Repeat-Dose Pharmacokinetics Study of NRL-1 in Epilepsy Subjects Under Seizure and Normal Conditions
Brief Title: Repeat-Dose Pharmacokinetics Study of NRL-1 in Epilepsy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurelis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAZ.001.04
Record Dates: First submitted 2016-03-17; First posted 2016-03-31 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-08

CONDITIONS: Acute Repetitive Seizures
Keywords: epilepsy; seizure
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Masking Description: open-label
Oversight: Data Monitoring Committee: No

ARMS (2):
- NRL-1 Ictal (Experimental): During the ictal or peri-ictal setting, a single intranasal dose of NRL-1 will be administered at either 5 mg, 10 mg, 15 mg, or 20 mg based on the subject's body weight.
  Interventions: Drug: NRL-1
- NRL-1 Inter-Ictal (Experimental): During the inter-ictal setting, a single intranasal dose of NRL-1 will be administered at either 5 mg, 10 mg, 15 mg, or 20 mg based on the subject's body weight.
  Interventions: Drug: NRL-1

INTERVENTIONS:
Drug: NRL-1
  Other Names: Intranasal diazepam

SUMMARY:
This study evaluates the pharmacokinetic and safety of NRL-1 in epilepsy subjects. Subjects will receive a single intranasal dose of NRL-1 of either 5 mg, 10 mg, 15 mg or 20 mg and will be based on the subject's body weight.

DETAILED DESCRIPTION:
Diazepam rectal gel (Diastat) is the only formulation of diazepam indicated for the management of selected, refractory patients with epilepsy on stable regimens of antiepileptic drugs (AEDs) who require intermittent use of diazepam to control bouts of increased seizure activity, i.e., Acute Repetitive Seizures (ARS).

A diazepam nasal spray is being developed for patients who experience ARS to provide an alternative more convenient and acceptable route of diazepam administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 6 and 65 years, inclusive.
2. Written informed consent to participate in the study.
3. Body mass index (BMI) not to exceed 35 kg/m², inclusive.
4. Subject has a clinical diagnosis of Epilepsy and, in the opinion of the Investigator, may need benzodiazepine intervention for seizure control.
5. Subjects having either partial or generalized Epilepsy with motor seizures or seizures with clear alteration of awareness are eligible for enrollment.
6. Female subjects of childbearing potential, defined as having a menstrual cycle and who are not surgically sterile or less than two (2) years postmenopausal, must complete a pregnancy screen and agree to utilize one of the following forms of contraception during the trial and for 21 days after the last dose of study drug: abstinence, hormonal (oral, transdermal, implant, or injection), barrier (condom, diaphragm with spermicide), intrauterine device (IUD), or vasectomized partner (six months minimum).
7. No clinically significant abnormal findings in the medical history, on the physical examination, ECG (corrected QT interval [QTcF] < 450 msec for males and QTcF < 470 msec for females), or clinical laboratory results during screening.
8. Subjects and caregivers must agree to return to the study site for all study visits and must be willing to comply with all required study procedures.

Exclusion Criteria:

1. Subject is undergoing intracranial EEG monitoring.
2. A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, severe seasonal or non-seasonal allergies, nasal polyps or any nasal passage abnormality that could interfere with nasal spray administration, or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
3. Subject has had significant traumatic injury, major surgery or open biopsy within 30 days prior to study screening.
4. Subjects with active major depression or a past suicide attempt documented on the Baseline/Screening C-SSRS. The children C-SSRS should be used for subjects age 6 to 11. The adult C-SSRS should be used for subjects 12 and greater years of age.
5. Any Suicidal Ideation of 3, 4, or 5 or any Suicidal Behavior in Lifetime using C-SSRS.
6. A history of allergic or adverse responses to diazepam or any comparable or similar product.
7. Subjects who (for whatever reason) have been on an abnormal diet (such as one that severely restricts specific basic food groups [e.g., ketogenic diet], limits calories [e.g., fast], and/or requires the use of daily supplements as a substitute for the foods typically eaten at mealtimes), during the four (4) weeks preceding the study.
8. Subjects who donated blood or plasma within 30 days of the first dose of study drug.
9. Participation in a clinical trial within 30 days prior to the first dose of study drug. Participation in an observational (non-interventional) study is not excluded as long as there are no scheduling conflicts with this study.
10. Inadequate or difficult venous access that may jeopardize the quality or timing of the PK samples.
11. Female subjects who are trying to conceive, are pregnant, or are lactating.
12. Positive serum pregnancy test (ß-hCG) at screening or urine pregnancy test prior to each administration of study drug for all women of childbearing potential.
13. Positive blood screen on subjects age 12 or greater for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HbSAg), or Hepatitis C, or a positive urine screen for alcohol, drugs of abuse, or cotinine. When marijuana was used for medical reasons in the opinion of the investigator, it is not considered as drug abuse and the patient can be enrolled even if the marijuana metabolites in the urine revealed as positive.
14. Treatment with phenobarbital or primidone within 30 days of the anticipated dosing visit (i.e., baseline).
15. Treatment with warfarin or dabigatran or other blood thinners within 30 days of the anticipated dosing visit (i.e., baseline).
16. Treatment with any diazepam containing products within 14 days of the anticipated dosing visit (i.e., baseline).
17. Use of nasal decongestants or nasal steroids within 7 days prior to the screening visit or during the study.
18. Subject does not have the flu, rhinitis or any other nasal condition that would impact absorption of intranasal diazepam.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Washington University School of Medicine, St Louis, Missouri
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospita, Memphis, Tennessee
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hogan RE, Tarquinio D, Sperling MR, Klein P, Miller I, Segal EB, Rabinowicz AL, Carrazana E. Pharmacokinetics and safety of VALTOCO (NRL-1; diazepam nasal spray) in patients with epilepsy during seizure (ictal/peri-ictal) and nonseizure (interictal) conditions: A phase 1, open-label study. Epilepsia. 2020 May;61(5):935-943. doi: 10.1111/epi.16506. Epub 2020 Apr 27. PMID 32338380

RESULTS

PARTICIPANT FLOW:
Groups:
- NRL-1: Single intranasal doses of NRL-1 (diazepam nasal spray) in epilepsy subjects during the ictal/peri-ictal period and single intranasal doses of NRL-1 (diazepam nasal spray) to the same subjects during the inter-ictal period.
Period: Overall Study
Arm/Group | NRL-1
Started | 57
Completed | 54
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | NRL-1
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 37
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (15.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 46
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Diazepam After Single Intranasal Doses of NRL-1 (Diazepam Nasal Spray) Administered to Epilepsy Subjects During the Ictal or Peri-ictal Period
Description: Evaluate the pharmacokinetics (PK), in terms of Cmax, of diazepam following a single intranasal dose of NRL-1 (diazepam nasal spray) administered to epilepsy subjects in the ictal or peri-ictal state (defined as either during or immediately following a seizure), where the seizure involved motor activity or alteration of awareness compared with the normal (non-seizing) state. The epileptic condition (ictal/peri-ictal, interictal) had minimal impact on diazepam nasal spray pharmacokinetics.
Time Frame: Blood samples were obtained at 0, 15, 30, and 45 minutes, and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, and 6 hours after dosing. If feasible, samples were drawn at 8 and 12 hours post-dose but were excluded from PK analysis.
Population: Of the 57 subjects who received NRL-1 and were included in the safety analysis dataset, there were 47 subjects per arm (82.5%) in the pharmacokinetic analysis dataset.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- NRL-1 ICTAL/PERI-ICTAL: NRL-1 ICTAL/PERI-ICTAL: This was a Phase 1, open-label, PK Study of Diazepam After Single Intranasal Doses of NRL-1 Administered to epilepsy Subjects During the Ictal or Peri-ictal Period.
- NRL-1 INTER-ICTAL: NRL-1 INTER-ICTAL: This was a Phase 1, open-label, PK Study of Diazepam After Single Intranasal Doses of NRL-1 Administered to epilepsy Subjects During the Inter-ictal Period.
Arm/Group | NRL-1 ICTAL/PERI-ICTAL | NRL-1 INTER-ICTAL
Number analyzed (Participants) | 47 | 47
ng/mL | 135 (88.6) | 153 (81.2)

2. Secondary Outcome: The AUC of Diazepam After Single Intranasal Doses of NRL-1 (Diazepam Nasal Spray) Administered to Epilepsy Subjects During the Ictal or Peri-ictal Period
Description: Evaluate the pharmacokinetics (PK), in terms of AUC, of diazepam following a single intranasal dose of NRL-1 (diazepam nasal spray) administered to epilepsy subjects in the ictal or peri-ictal state (defined as either during or immediately following a seizure), where the seizure involved motor activity or alteration of awareness compared with the normal (non-seizing) state. The epileptic condition (ictal/peri-ictal, interictal) had minimal impact on diazepam nasal spray pharmacokinetics.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | NRL-1 ICTAL/PERI-ICTAL | NRL-1 INTER-ICTAL
Number analyzed (Participants) | 47 | 47
ng*hr/mL | 435 (85.0) | 502 (78.1)

ADVERSE EVENTS:
Time Frame: Up to 65 days
Groups:
- NRL-1: A single intranasal dose of NRL-1 will be administered at either 5 mg, 10 mg, 15 mg, or 20 mg based on the subject's body weight.
  NRL-1
Arm/Group | NRL-1
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 1/57
Other Adverse Events (participants affected / at risk) | 9/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRL-1 (N=57)
Recurrent seizures (Nervous system disorders) | 1 (1)
Static encephalopathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRL-1 (N=57)
Dysgeusia (Nervous system disorders) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT02724423/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT02724423/SAP_001.pdf